CLINICAL TRIAL: NCT04097210
Title: When Triage is Insufficient - the Benefit of Bedside CRP Within Ambulance Care
Brief Title: Decision-making - the Benefit of Bedside CRP Within Ambulance Care
Acronym: Q-CRP
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Marja Mäkinen, PhD, principal investigator, Helsinki University Central Hospital
Other Study IDs: HUS 329/13/3/02/2015
Record Dates: First submitted 2018-11-26; First posted 2019-09-20 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2018-11

CONDITIONS: Critical Illness
Keywords: Q-CRP; lactate; suPAR; POC; ambulance
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No biospecimen banking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: POC

SUMMARY:
Patients with degreased (DGC) for ambiguous reasons receive low triage priority. Their death risk is triple. Tools are needed to identify the critically ill patients from this group. The triage used today is not effective. The bedside point-of-care measurements are CRP, lactate acid and suPAR (Soluble Urokinase Plasminogen Activator Receptor). Elevated values associate with the probability of critical illness and predict a risk of death.

DETAILED DESCRIPTION:
Purpose: To improve identification and proper prioritization of patients with non-specific symptoms prehospitally, we intend to investigate whether Q-CRP, a rapid test for CRP, correlates with time-critical states in the above-mentioned patient group alone or together with CRP, lactate and suPAR. The primary endpoint is need for hospital care.

Material: Patients over 18 years who exhibit non-specific symptoms and transported to the emergency room.

Method: In patients with unspecified conditions, defined according to the inclusion template, a venous blood sample was taken prehospitally at the scene by the EMS.

Analysis: Significance tests and regression analyzes with 95% CI were used. The diagnostic accuracy of Q-CRP, lactate, suPAR and combinations thereof were compared with optimal boundary values.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years who exhibit non-specific symptoms and transported to the emergency room.

Exclusion Criteria:

* Abnormal vitals

Ages: 16 Years to 104 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with degreased condition (DGC) over 18 years who exhibit non-specific symptoms and transported to the emergency room.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with high suPAR level | 24 hours
  A high suPAR level, e.g. above 6 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Maaret Castrén, Professor, Study Director — Helsinki University Central Hospital; Johanna Kaartinen, PhD, Principal Investigator — Helsinki University Central Hospital